CLINICAL TRIAL: NCT00873522
Title: Microbiology and Clinical Outcome of Community Acquired Pneumonia and Health-Care-Associated Pneumonia in Taiwan: a Multi-Center Study
Brief Title: Microbiology and Clinical Outcome of Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Chieh-Liang Wu, Department of Respiratory Therapy, Taichung Veterans General Hospital
Other Study IDs: C08012
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Pneumonia
Keywords: pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Community acquired pneumonia
- Health-Care-Associated pneumonia

SUMMARY:
1. BACKGROUND

   Pneumonia occurring outside of the hospital setting is regarded as community acquired pneumonia. However, pneumonia occurring in non-hospital long-term care facilities constituted a distinct type of pneumonia from CAP. Kollef et al has justified health care associated pneumonia (HCAP) as a new category of pneumonia [1]. The HCAP patients are associated with severe disease, higher mortality rate, and greater length of stay and increased cost [1]. HCAP are often at risk for multi-drug resistant bacterial pathogens such as Pseudomonas aeruginosa, extended-spectrum beta-lactamase Klebsiella pneumoniae, Acinetobacter baumannii, and methicillin-resistant S. aureus (MRSA) [2].

   Health care facilities have not been defined in Taiwan. Respiratory care ward (RCW) is a special unit to take care long-term ventilatory dependent patients in Taiwan. Some of the patients get pneumonia and are referred back to medical centers. Besides, community-acquired P. aeruginosa, Acinetobacter baumannii or MRSA have been reported [3-8]. Therefore, the core-organisms of HCAP in Taiwan might be multi-drug resistant and the causes of inadequate initial antibiotics treatment. The common pathogens were also unknown.

   Till now, there are no data about the pathogens of HCAP in Taiwan. We define the health-care facilities and initiate a retrospective study to characterize the microbiology and clinical outcome of Community acquired pneumonia and Health-Care-Associated pneumonia in Taiwan. Further analysis will perform to confirm the differences between CAP an HCAP in Taiwan.
2. Objectives:

   I. To characterize CAP and HCAP i. Microbiological epidemiology ii. Disease severity: PSI iii. Outcome : length of stay, mortality , antimicrobial susceptibility and treatment outcomes II. To characterize HCAP from RCW i. Microbiological epidemiology ii. Disease severity: PSI iii. Outcome : length of stay, mortality
3. Study design:

This is a retrospective multi-center cohort study to characterize microbiology, and clinical outcomes in Taiwan.

Data sources: CAP or HCAP registered in 4 medical centers from Jan 1 2007 to Dec. 31 2007. (2 in north Taiwan, 1 in central Taiwan, 1 in south Taiwan) Expected case number: 800 HCAP and 1800 CAP

DETAILED DESCRIPTION:
BACKGROUND

Pneumonia occurring outside of the hospital setting is regarded as community acquired pneumonia. However, pneumonia occurring in non-hospital long-term care facilities constituted a distinct type of pneumonia from CAP. Kollef et al has justified health care associated pneumonia (HCAP) as a new category of pneumonia . The HCAP patients are associated with severe disease, higher mortality rate, and greater length of stay and increased cost - HCAP are often at risk for multi-drug resistant bacterial pathogens such as Pseudomonas aeruginosa, extended-spectrum beta-lactamase Klebsiella pneumoniae, Acinetobacter baumannii, and methicillin-resistant S. aureus (MRSA) Health care facilities have not been defined in Taiwan. Respiratory care ward (RCW) is a special unit to take care long-term ventilatory dependent patients in Taiwan. Some of the patients get pneumonia and are referred back to medical centers. Besides, community-acquired P. aeruginosa, Acinetobacter baumannii or MRSA have been reported [3-8]. Therefore, the core-organisms of HCAP in Taiwan might be multi-drug resistant and the causes of inadequate initial antibiotics treatment. The common pathogens were also unknown.

Till now, there are no data about the pathogens of HCAP in Taiwan. We define the health-care facilities and initiate a retrospective study to characterize the microbiology and clinical outcome of Community acquired pneumonia and Health-Care-Associated pneumonia in Taiwan. Further analysis will perform to confirm the differences between CAP an HCAP in Taiwan.

Objectives:

* To characterize CAP and HCAP
* Microbiological epidemiology
* Disease severity: PSI
* Outcome : length of stay, mortality , antimicrobial susceptibility and treatment outcomes
* Microbiological epidemiology
* Disease severity: PSI
* Outcome : length of stay, mortality

Study design:

This is a retrospective multi-center cohort study to characterize microbiology, and clinical outcomes in Taiwan.

Data sources: CAP or HCAP registered in 4 medical centers from Jan 1 2007 to Dec. 31 2007. (2 in north Taiwan, 1 in central Taiwan, 1 in south Taiwan) Expected case number: 800 HCAP and 1800 CAP

Study population:

Those adult patients (age ≥ 18 y/o) met the criteria of pneumonia are evaluated. The patients are enrolled if they meet the following criteria.

The diagnosis of pneumonia is established within 48h of hospitalization (including time of emergency room).

Pneumonia is defined as clinical suspicion of pneumonia (cough, short of breath, expectorant) with new-onset pulmonary infiltrates plus at least one of the following criteria:

* Fever (≥38.3 C) or hypothermia (<36.0 C) (axillary temp - 0.5)
* Leukocytosis (increase of total WBC > 10,000/cumm); or leukopenia (<4000/cumm) or band > 10%
* Purulent airway secretion (tracheal aspirates, or sputum)

Etiology diagnosis

* Specimens obtained within 72h (sputum, tracheal aspirate, BAL, pleural effusion or blood)
* Urine antigen test for legionella or Streptococcus at the onset of pneumonia
* Paired serology (at admission and within 4th to 8th weeks)
* virus culture
* Definition of definite pathogen: [9](Resp Med 2005;1079)
* Blood culture is accepted if the same microorganism is identified in a respiratory specimens and no other source for the positive blood culture could be identified.
* The isolate is cultured from pleural effusion.
* ≥ 4 x fold risk in IgG antibody titer to L. pneumoniae, C. pneumoniae or to any of respiratory virus antigens tested or a seroconversion of antibodies to M. pneumoniae based on manufacture's criteria.
* M. pneumoniae IgM (+), L. pneumoniae ( IgG higher above 1:128) or C. pneumoniae ( high above 1:256) are also defined as definite pathogens.
* Detection of L. pneumoniae antigen in urine
* Detection of S. pneumoniae antigen in urine or isolation of S. pneumoniae from purulent sputum
* Bronchoscope guided study: BAL > 104/cfu, PSB > 103/cfu
* Sputum or BAL revealing Pneumocystic carinii, Mycobacterium tuberculosis, Cryptococcus neoformans
* Growth of fungi in the respiratory samples is considered diagnostic only in the presence of a concomitant positive blood culture growing the same microorganism (candida, Aspergillosis)

Probable pathogens:

* Pathogen was confirmed by the isolatioin of a predominant organism from sputum or endotracheal aspirate

Comorbidity:

* Neoplastic disease
* Any cancer except basal or squamous cell ca of the skin that was active at the time of presentation or diagnosed within one year of presentation
* Liver disease
* A clinical or histologic diagnosis of cirrhosis or another form of chronic liver disease such as chronic active hepatitis
* Cardiac comorbid illness:
* Systolic or diastolic ventricular dysfunction documented by history, physical examination, chest radiograph, echocardiogram, multiple gated acquisition scan or left ventriculogram (congestive heart failure New York heart association class III to IV)
* Disorders of the central nervous systems
* A clinical diagnosis of stroke or transient ischemic attack or stroke documented by MRI or CT scan
* Presence of symptomatic acute or chronic vascular or nonvascular encephalopathy, dementia, parkinsonism, motor neuron disease etc

Renal:

* A history of chronic renal disease or abnormal blood urea nitrogen and creatinine concentration documented in the medical record (Cr >2mg/dL)
* Pulmonary:

treatment for asthma, or COPD, or presence of interstitial lung disease, bronchiectasis, tuberculosis,

* DM

Lung cancer:

* Lung cancer active at the time of presentation or requiring anti-neoplastic treatment within the preceding one year.
* Autoimmune disease
* Treatment for RA, SLE, polymyositis, dermatomyositis etc
* Having an immunocompromised state
* equivalent to > daily prednisolone 5mg or > prednisolone 150 mg / month
* other immunosuppressive medications (cyclophosphamide, cyclosporine etc)
* s/p organ transplantation

Definition of clinical items:

Altered mental status: disorientation with respect to person, place or time that is not known to be chronic, stupor, or coma

* Neutropenia:

  * neutropenia with absolute neutrophil count < 1000
  * smoking (pack year)
  * current smoker
  * exsmoker (quitting for > 6 months)
  * non-smoker (never smoking)
* Septic shock: a persistent arterial hypotension in a septic patient.
* Hypotension is defined by a systolic arterial pressure < 90mmHg or Mean arterial pressure < 60mmHg after adequate volume resuscitation (>5000 cc fluid resuscitation/day) or vasopressor (dopamine > 5mcg/kg/h) to maintain blood pressure.
* Acute respiratory failure: need mechanical ventilation support intubation and MV support only non-invasive mechanical ventilator
* ICU admission: admission to ICU during hospitalization
* Length of ICU: days staying in ICU
* Hospital days: days staying in the hospital (from ER to hospital discharge) discharge status
* mortality (including AAD with impending death)
* survival
* without MV (invasive and non-invasive MV)
* tracheostomy
* ventilator dependent
* Residence after discharge
* Home, nursing home, RCW, others
* Organ failure:
* Respiratory failure（PaO2／FiO2<300 )
* Acute renal failure（Cr>2.0 or Cr increase>0.5 ㎎/dl )
* Acute liver failure（Total bilirubin>4 ㎎/dl )、
* Coagulopathy（INR>1.5 time or aPTT>60 seconds )
* Thrombocytopenia（Platelets <100000／CUMM ）

All parameters required for the calculation of PSI (Pneumonia Severity Index, appendix) at baseline will be collected.

Definition of appropriateness of Empirical therapy Empirical antibiotic therapy is defined as antibiotic given during the first 48 hours for pneumonia. The appropriateness of antibiotic therapy will be analyzed only for cases with causative organism (probably and definite organisms) identified. Inadequacy therapy is defined as administration of an antibiotic to which the isolated pathogen was resistant according to the subsequent antimicrobial susceptibility results or the absence of antimicrobial agents to cover the identified pathogen(s). In addition, patients with aspiration pneumonia (Aspiration pneumonia are defined as witnessed aspiration pneumonia and food or material noted in the upper or lower airways) who had not received agents with anti-anaerobic coverage will be considered inappropriate.

Definition of Treatment outcomes

In addition to collecting microbiological response, clinical response data will be used for all patients. Success/favorable clinical response will be defined as all or most of pretreatment signs and symptoms of the index infection have resolved or improved (e.g.: TPR shift toward normal) and no additional antibiotic therapy or switching of regimen was required. While failure will be defined as no apparent response to therapy; persistence or progression of most/all pre-therapy signs and symptoms and additional antibiotic therapy or switching of regimen was documented.

Cases will be classified as "Indeterminate" when no sufficient data is available to permit evaluation of microbiological or clinical outcome or patient's underlying medical condition is too complicated to precluded classification as a success or failure.

Data collection and analysis plan

Data from all sites will be pooled and combined. Statistical analyses will be conducted with the use of SAS software, version 8.2 (SAS Institute Inc., Cary, NC, USA). Data will also be presented as mean +/-SD for continuous variables and proportions for categories variables. The patient demographics and baseline characteristics will be tabulated. The distribution of comorbidities, disease severity, causative organisms, clinical condition and outcomes will be summarized and analyzed. To detect the significant differences between groups, Chi-square tests or Fisher exact test for categorical variables, and the two-tailed t test or Mann-Whitney test for continuous variables will be employed, when appropriate. Statistical significance will be established at alpha =0.05. Reported P values will be two-sided.

ELIGIBILITY:
Inclusion Criteria:

CAP criteria:

* Those pneumonia patients have not been admitted within 14 days before diagnosing pneumonia.
* Those pneumonia patients are not met the criteria of HCAP criteria as stated below.

HCAP criteria:

* Regular hemodialysis, peritoneal dialysis or infusion therapy (ex TPN, repeated blood transfusion etc ) at a hospital or hemodialysis clinic.
* Receive radiation therapy or chemotherapy at out-patient clinics within 90 days
* to be admitted to an acute care hospital for two or more days within 90 days before the onset of pneumonia
* Resided in a nursing home or long-term care

Exclusion Criteria:

* The patients with HAP: pneumonia developed two days after admission or within 14 days after discharge (except RCW)
* VAP: HAP and with mechanical ventilation for at least 48h (except RCW patients)
* HIV positive with a CD4+ < 200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those adult patients (age ≥ 18 y/o) met the criteria of pneumonia are evaluated. The patients are enrolled if they meet the following criteria [9] .
  * The diagnosis of pneumonia is established within 48h of hospitalization (including time of emergency room).
  * Pneumonia is defined as clinical suspicion of pneumonia (cough, short of breath, expectorant) with new-onset pulmonary infiltrates plus at least one of the following criteria:
    * Fever (≥38.3C) or hypothermia (<36.0C) (axillary temp - 0.5)
    * Leukocytosis (increase of total WBC > 10,000/cumm); or leukopenia (<4000/cumm) or band > 10%
    * Purulent airway secretion (tracheal aspirates, or sputum)
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Success/favorable clinical response after treatment for pneumonia | weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Liang Wu, MD, Principal Investigator — Department of Respiratory Therapy, Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan